CLINICAL TRIAL: NCT00818987
Title: A Multicentre Prospective Randomized Control Trial on the Treatment of Three and Four Part Proximal Humerus Fractures in Patients 70 Years and Older: Comparing Open Reduction and Internal Fixation With Non Operative Treatment
Brief Title: Operative Versus Non Operative Treatment of Proximal Humerus (Shoulder Joint) Fractures
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Pierre Guy, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-02149
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: 3 and 4 Part Proximal Humerus Fractures
Keywords: Operative; Non operative
MeSH Terms: interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative (Other): Treatment arm - intervention = Open Reduction Internal Fixation or Reduction & Immobilization
  Interventions: Other: Open reduction internal fixation; reduction and immobilization
- Non Operative (No Intervention): Placebo arm

INTERVENTIONS:
Other: Open reduction internal fixation; reduction and immobilization
  Arms: Operative

SUMMARY:
To determine if operative treatment of non operative management of these fractures is best. Hypothesis: There is no difference in functional outcome between operative and non-operatively treated 3- and 4-part proximal humerus fractures at one year's time.

DETAILED DESCRIPTION:
Participants of 70 years of age or older who have been medically assessed as 'fit for surgery' are randomly (like flipping a coin) to either operative or non operative management of their injury. Clinical follow-up including x-rays, and physical assessment of injured shoulder, and outcomes questionnaires will be used to determine which if either resulted in the best outcome.

ELIGIBILITY:
Inclusion Criteria:

* Proximal humerus fracture patients

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-05 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measurement will be the patients' functional shoulder scores as measured by the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire | 1 year

SECONDARY OUTCOMES:
Functional and mental status instruments (i.e. SF-36/EQ-5D) used to assess the patient's health-related quality of life;, re-operation rates; and the time required to return to pre-injury level of independence | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Guy, MDCM, MBA, FRCS(C), Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196